CLINICAL TRIAL: NCT05262621
Title: Effects of Music Intervention Combined With Progressive Muscle Relaxation on Anxiety, Depression and Quality of Life in Breast and Gynaecological Cancer Patients Receiving Chemotherapy: A Randomized Controlled Trial
Brief Title: Effects of Music Intervention Combined With Progressive Muscle Relaxation in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Nethersole School of Nursing (Other)
Responsible Party: Principal Investigator, Khanh Thi Nguyen, Principal Investigator, The Nethersole School of Nursing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TheNethersole
Record Dates: First submitted 2022-02-09; First posted 2022-03-02 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Cancer
Keywords: music intervention; progressive muscle relaxation; anxiety; depression; quality of life; chemotherapy; beast cancer; gynaecology cancer
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression | interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: The research assistants who assess outcome data, data entry and analysis will be blinded to avoid the risk of assessor bias. The assistants will not participate in any other stage of implementing the program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music intervention combined with progressive muscle relaxation (Experimental): Music intervention combined with progressive muscle relaxation.
  Interventions: Other: progressive muscle relaxation; Other: Listening to relaxing music once/day
- Control group (No Intervention): no music therapy will be done.

INTERVENTIONS:
Other: progressive muscle relaxation — Practice muscle relaxation for 20 minutes once/a day
  Arms: Music intervention combined with progressive muscle relaxation
Other: Listening to relaxing music once/day — Right after practising progressive muscle relaxation, the participants will listen to relaxing music for 20 minutes
  Arms: Music intervention combined with progressive muscle relaxation

SUMMARY:
Study design A 2-arm, assessor-blinded randomised controlled trial will be conducted. The design will follow the Standard Protocol Items Recommendations for Interventional Trials (SPIRIT)

DETAILED DESCRIPTION:
Aim: To assess the effect of MCP on anxiety, depression and QoL of BGC patients receiving chemotherapy.

Objectives

* To assess the effect of MCP on the anxiety of BGC patients receiving chemotherapy.
* To assess the effect of MCP on depression of BGC patients receiving chemotherapy.
* To assess the effect of MCP on QoL and patients' satisfaction of BGC patients receiving chemotherapy.
* To determine whether stress level, coping and coping styles mediate the intervention effect on anxiety, depression and QoL.

Hypothesis

* The participants receiving MCP will have a significantly lower level of anxiety compared to the control group.
* The participants receiving MCP will have a significantly lower level of depression compared to the control group.
* The participants receiving MCP will have significantly higher QoL scores and levels of satisfaction with care service compared to the control group.
* Stress level, coping will mediate the intervention on target outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women with breast or gynaecological cancer are 18 years of age or older, and are independent legally to sign the consent form.
* Living with family and having an adult family member agree to participate in the meeting part of the program.
* Had been informed the cancer diagnosis
* Have Karnofsky score (Mor et al., 1984) ≥ 80 ( to be able to self-practice MCP)
* Can communicate, read and write in Vietnamese
* Have a device such as a smartphone, MP3 to keep the audio file (to self-practice MCP at home)
* Consent to join the study

Exclusion Criteria:

* The patients cannot understand the study procedures
* Have mental health illness, deafness, blindness
* Have not been aware of their cancer or the purpose of chemotherapy
* Be participating in other studies related to psychological issues
* Be receiving anxiety or depression treatment.
* Be participating in relaxation therapy such as yoga, meditation, mindfulness, PMR...
* Have a potential treatment (eg. surgery) or personal plans that will prevent them from practising daily during the 6 weeks of the intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline anxiety at 3 weeks and 6 weeks | ebaseline, T1 after 3 weeks, T2 after 6 weeks
  it will be measured using the short form of the Depression Anxiety Stress Scale (DASS-21). It includes 7 items for anxiety (DASS21-A). A 4-point Likert-type scale ranging from 0 to 3 was designed for each item, and the scores will need to be multiplied by 2 to calculate the final score. Thus, the anxiety score can range from 0 to 42. The higher the score is the more severe anxiety. The score of 0-7 is normal, 8-9 mild, 10-14 moderate, 15-19 severe, +20 extremely severe.
Change from baseline depression at 3 weeks and 6 weeks | baseline, T1 after 3 weeks, T2 after 6 weeks
  it will be measured using the short form of the Depression Anxiety Stress Scale (DASS-21). It includes 7 items for depression (DASS21-D). A 4-point Likert-type scale ranging from 0 to 3 was designed on each item, and the scores will need to be multiplied by 2 to calculate the final score. Thus, the depression score can range from 0 to 42. The higher the score is the more severe depression. The score of 0-9 is normal, 10-13 mild, 14-20 moderate, 21-27 severe, +28 extremely severe.

SECONDARY OUTCOMES:
Change from baseline stress at 3 weeks and 6 weeks | baseline, T1 after 3 weeks, T2 after 6 weeks
  it will be measured using the short form of the Depression Anxiety Stress Scale (DASS-21). It includes 7 items for stress (DASS21-S). A 4-point Likert-type scale ranging from 0 to 3 was designed for each item, and the scores will need to be multiplied by 2 to calculate the final score. Thus, the stress score can range from 0 to 42. The higher the score is the more severe stress. The score of 0-14 is normal, 15-18 mild, 19-25 moderate, 26-33 severe, +34 extremely severe.
Change from baseline coping styles at 3 weeks and 6 weeks | baseline, T1 after 3 weeks, T2 after 6 weeks
  Coping will be measured using Brief COPE. The Brief-COPE is a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event.The scale can determine someone's primary coping styles with scores on the following three subscale:
  Problem-Focussed Coping, Emotion-Focussed Coping, Avoidant Coping.A 4-point Likert-type scale ranging from 1 to 4 was designed on each item.
Change from baseline quality of life at 3 weeks and 6 weeks | baseline, T1 after 3 weeks, T2 after 6 weeks
  coping will be measured using FACT-G.It evaluates in functional scales on Social/family well-being (SWB); Emotional well-being (EWB) and Functional well-being (FWB). Each item is scored in one of five categories of 0-4, with 'Not at all', 'A little bit', 'some what', 'Quite a bit' 'Very much'. The higher the score is the better quality of life." The possible range of scores is from 0 to 112.
Change from baseline satisfaction of nursing care at 3 weeks | baseline, T1 after 3 weeks,
  satisfaction of nursing care will be measured using numerical rating scale.(0-10) from 0 = completely dissatisfied with the care to 10 = completely satisfied with the care.

CONTACTS AND LOCATIONS:
Overall Officials: Khanh Thi Nguyen, master, Principal Investigator — The Nethersole School of Nursing, The Chinese University of Hong Kong
Locations (1):
- Vietnam National Cancer Institute, Hanoi Oncology Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen KT, Chan DNS, Cheung AT, Hoang HTX, Truong AT, Chow KM, Choi KC, Chan CWH. Randomised controlled trial of music listening combined with progressive muscle relaxation for mood management in women receiving chemotherapy for cancer. Support Care Cancer. 2025 Mar 4;33(3):245. doi: 10.1007/s00520-025-09281-4. PMID 40035884
- [Derived] Nguyen KT, Hoang HTX, Bui QV, Chan DNS, Choi KC, Chan CWH. Effects of music intervention combined with progressive muscle relaxation on anxiety, depression, stress and quality of life among women with cancer receiving chemotherapy: A pilot randomized controlled trial. PLoS One. 2023 Nov 3;18(11):e0293060. doi: 10.1371/journal.pone.0293060. eCollection 2023. PMID 37922279